CLINICAL TRIAL: NCT07258771
Title: Acute Severe Ulcerative Colitis- Upadacitinib Combined With Corticosteroids vs Corticosteroid Monotherapy Induction While Transitioning Away From the Emergency Setting (ACUTE): A Phase IV, Single Center, Partially Blinded, Randomized Study
Brief Title: Upadacitinib Combined With Corticosteroids vs Corticosteroid Monotherapy Induction for Inpatients and Outpatients With Acute Severe Ulcerative Colitis
Acronym: ACUTE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Berinstein, Jeffrey (Other)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor-Investigator, Berinstein, Jeffrey, Assistant Professor of Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00266952
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis Acute
Keywords: Acute Severe Ulcerative Colitis; Inpatient; Outpatient; Optimal sequence; Upadacitinib; Corticosteroids
MeSH Terms: interventions — upadacitinib; Methylprednisolone Hemisuccinate; Prednisone

STUDY DESIGN:
Intervention Model Description: This study will implement a partially double-blind design, where the inpatient/outpatient treatment team, investigators, and participants will be blinded to the assigned treatment throughout the acute induction phase. If rescue therapy is initiated the outpatient or inpatient group the participants will be unblinded. For participants in the inpatient cohort that do not receive rescue therapy, treatment assignment will be unblinded once participants are discharged to guide the choice of maintenance therapy for those in the corticosteroid arm. Additionally, participants in the outpatient cohort will be unblinded on Day 5 to facilitate the selection of maintenance therapy for the corticosteroid arm. Following these specified unblinding events, the remainder of the trial, including the post-acute induction and maintenance phases, will be open label with no further blinding.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Upadacitinib plus steroids-Outpatient cohort (Experimental): This will include patients who meet acute severe ulcerative colitis criteria who are seen in clinic, that contact the clinic, or are sent to the ambulatory, diagnostic and treatment unit (ADTU) without requiring an admission to the hospital.
  Participants will receive upadacitinib 45mg and hospital dose steroids (IV Methylprednisolone 60mg in an infusion center or ADTU or PO Prednisone 75mg) up to Day 5. If the participant's condition does not improve or if it worsens after 3 days from starting assigned treatment, the participant will be unblinded and put on "rescue therapy". Unrescued participants will be unblinded on Day 5 when the Acute Induction Phase is complete.
  Upon completion of the Acute Induction Phase, participants will receive upadacitinib 45 mg for 8 weeks concomitant with a 2-week prednisone course.
  Upadacitinib therapy may continue through week 48, with dosage (45 mg, 30 mg, or 15 mg) titrated based on clinical symptoms and inflammatory biomarkers.
  Interventions: Drug: Oral Upadacitinib; Drug: Intravenous Methylprednisolone; Drug: Oral prednisolone Taper; Drug: Oral Prednisone - Hospital Dose Steroids
- Steroids plus Upadacitinib Placebo-Outpatient cohort (Active Comparator): This will include patients who meet acute severe ulcerative colitis criteria who are seen in clinic, that contact the clinic, or are sent to the ambulatory, diagnostic and treatment unit (ADTU) without requiring an admission to the hospital.
  Participants will receive upadacitinib placebo and hospital dose steroids (IV Methylprednisolone 60mg in an infusion center or ADTU or PO Prednisone 75mg) up to Day 5. If the participant's condition does not improve or if it worsens after 3 days from starting assigned treatment, the participant will be unblinded and put on "rescue therapy".
  Unrescued participants will be unblinded on Day 5 to guide selection of maintenance therapy. Upon completion of the Acute Induction Phase, participants will receive taper prednisone by 5mg per week starting at 40mg with maintenance therapy initiation per usual care.
  Interventions: Drug: Intravenous Methylprednisolone; Drug: Oral Upadacitinib Placebo; Drug: Oral prednisolone Taper; Drug: Oral Prednisone - Hospital Dose Steroids
- Upadacitinib plus steroids- Inpatient cohort (Experimental): This will include patients seen in the Emergency Department or who are hospitalized. Participants will receive upadacitinib 45mg and hospital dose steroids (IV Methylprednisolone 60mg) until they are discharged. If the participant's condition does not improve or if it worsens after 3 days from starting assigned treatment, the participant will be unblinded and put on "rescue therapy". Unrescued participants will be unblinded as soon as participants are discharged (completion of the Acute Induction Phase).
  Upon completion of the Acute Induction Phase, participants will receive upadacitinib 45 mg for 8 weeks concomitant with a 2-week prednisone course.
  Upadacitinib therapy may continue through week 48, with dosage (45 mg, 30 mg, or 15 mg) titrated based on clinical symptoms and inflammatory biomarkers.
  Interventions: Drug: Oral Upadacitinib; Drug: Intravenous Methylprednisolone; Drug: Oral prednisolone Taper
- Steroids plus Upadacitinib Placebo- Inpatient cohort (Active Comparator): This will include patients seen in the Emergency Department or who are hospitalized. Participants will receive upadacitinib placebo and hospital dose steroids (IV Methylprednisolone 60mg) until they are discharged. If the participant's condition does not improve or if it worsens after 3 days from starting assigned treatment, the participant will be unblinded and put on "rescue therapy". Unrescued participants will be unblinded as soon as participants are discharged (completion of the Acute Induction Phase) to guide maintenance therapy selection (outside of the trial protocol).
  Upon completion of the Acute Induction Phase, participants will taper prednisone by 5mg per week starting at 40mg with maintenance therapy initiation per usual care.
  Interventions: Drug: Intravenous Methylprednisolone; Drug: Oral Upadacitinib Placebo; Drug: Oral prednisolone Taper

INTERVENTIONS:
Drug: Oral Upadacitinib — Doses start at 45milligrams (mg) during acute induction and post-acute induction phase (total of 8 weeks).
  During the Dose Optimization Maintenance Phase, unrescued participants not undergoing colectomy will continue upadacitinib therapy through week 48, with dosage (45 mg, 30 mg, or 15 mg) titrated based on clinical symptoms and inflammatory biomarkers.
  Other Names: Rinvoq
  Arms: Upadacitinib plus steroids- Inpatient cohort; Upadacitinib plus steroids-Outpatient cohort
Drug: Intravenous Methylprednisolone — Intravenous (IV) given 60mg daily (in divided or full doses). Inpatients will receive this in the hospital. Outpatient participants can get this at an infusion center.
  Following completion of the Acute Induction Phase (inpatient cohort: 0-10 days ending at discharge; outpatient cohort: 5 days), participants will be placed on a tapering dose of prednisone.
  Other Names: Solumedrol
Drug: Oral Upadacitinib Placebo — The placebo will be discontinued at discharge for the inpatient cohort and after day 5 for the outpatient cohort.
  Other Names: Placebo
  Arms: Steroids plus Upadacitinib Placebo- Inpatient cohort; Steroids plus Upadacitinib Placebo-Outpatient cohort
Drug: Oral prednisolone Taper — Following completion of the Acute Induction Phase (inpatient cohort: 0-10 days ending at discharge; outpatient cohort: 5 days), participants will be placed on a tapering dose of prednisone.
  Participants randomized to the corticosteroid arm will be placed on prednisone at a dose 40mg to be tapered by 5mg/week.
  Participants randomized to the upadacitinib and corticosteroid arm will be placed on 2 weeks of prednisone (40mg x 2 days, 30mg x 2 days, 25mg x 2 days, 20mg x 2 days, 15mg x 2 days, 10mg x 2 days, and 5mg x 2 days).
  Other Names: Prednisone
Drug: Oral Prednisone - Hospital Dose Steroids — Oral Prednisone 75mg daily can be given for 5 days to participants enrolled in the Outpatient Cohort as an alternative to getting IV methylprednisolone 60mg in an infusion center. Following completion of the Acute Induction Phase, participants will be placed on a tapering dose of prednisone.
  Other Names: prednisone
  Arms: Steroids plus Upadacitinib Placebo-Outpatient cohort; Upadacitinib plus steroids-Outpatient cohort

SUMMARY:
This trial is being conducted to learn more about the optimal sequence of various medications in the management of acute severe ulcerative colitis (ASUC).

This research is studying multiple drugs already approved by the Food and Drug Administration (FDA). The goal of this study is to test the early efficacy and safety of upadacitinib (Rinvoq) and corticosteroids compared to corticosteroids alone as induction therapy for both inpatients and outpatients with ASUC.

DETAILED DESCRIPTION:
This study will have four phases: eligibility assessment, the acute induction phase (inpatient 0-10 days, outpatient 5 days), post-acute induction phase (end of acute induction phase to day 56 (week 8)), and maintenance phase (week 8-week 48).

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 to 75 years of age at the time of consent
* Diagnosis of ulcerative colitis (verified by a typical clinical history as well as characteristic appearance on endoscopy and histology)
* Meeting the following definition of acute severe ulcerative colitis as defined as having ≥ 6 bowel movements per day with visible blood in the 7 days prior to Day 0 plus at least one of the following:

  i. Temperature > 37.8 Celsius(C) per patient report or documented in Electronic Health Record (EHR) in the 7 days prior to Day 0.

ii. Pulse ≥ 90 beats per minute (BPM) per patient report or documented in EHR iin the 7 days prior to Day 0 iii. Hemoglobin ≤ 10.5 grams per deciliter (g/dL) in the 7 days prior to Day 0 iv. Erythrocyte sedimentation rate ≥ 30 millimeters per hour (mm/h) in the 7 days prior to Day 0 v. C-reactive protein ≥ 3.0mg/dL in the 7 days prior to Day 0 vi. Fecal calprotectin >782 Milligrams per kilogram (mg/kg) in the 7 days prior to consent.

vii. Oral corticosteroid use for ≥ 7 days in the month prior to consent at a dose equivalent to ≥ 20 milligrams per day (mg/day)

* For a person of reproductive/childbearing potential (i.e., presence of intact ovaries and fallopian tubes and are considered premenopausal by standard assessment), a negative lab-based (serum/urine) pregnancy test is required.
* For a person of reproductive potential (i.e., presence of intact ovaries and fallopian tubes) and has childbearing potential, intent to use at least one effective method of birth control from study Day 0 through the end of blinding or at least 30 days after the last dose of upadacitinib or week 48, whichever occurs most recently. A person without reproductive or childbearing potential does not require an intent to use effective birth control.
* Participants enrolled in the outpatient cohort must be under the care of an outpatient gastroenterologist affiliated with the University of Michigan.
* Ability to take oral medication and be willing to adhere to the study intervention regimen.
* Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, daily bowel movement symptoms surveys, and other study procedures.
* Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* On IV corticosteroids for > 72 hours immediately prior to enrollment continuously (at any institution) which is equivalent to a cumulative dose of 180mg of IV Methylprednisolone in the 3 days prior to enrollment.
* Patients with a prior exposure upadacitinib. Previous exposure to other Janus kinase (JAK) inhibitors (e.g., tofacitinib, baricitinib, or filgotinib) are permissible.
* History of clinically significant (per investigator's judgment) drug or alcohol abuse within the last 6 months prior to Baseline. (Note: A Urine Drug Screen does not need to be performed).
* A history of two or more prior episodes of herpes zoster, or one or more episodes of disseminated herpes zoster.
* Patients with ongoing severe active infection (as determined by the study team) per investigator. Patients with active serious infection(s) requiring treatment with intravenous anti-infectives or oral/intramuscular anti-infectives may consider infectious disease clearance.
* Active tuberculosis (TB) or untreated latent TB as described in the protocol.
* In participants that tested positive for Coronavirus disease 2019 (COVID-19), at least 5 days must have passed between a COVID-19 positive test result and the baseline visit of asymptomatic participants. Participants with mild/moderate COVID-19 infection can be enrolled if fever is resolved without use of antipyretics for 24 hours and other symptoms improved, or if 5 days have passed since the COVID-19 positive test result (whichever comes last). Participants may be rescreened if deemed appropriate by the investigator based upon the participant's health status.
* Recent (within past 6 months) cerebrovascular accident, myocardial infarction, coronary stenting, or aorto-coronary bypass surgery.
* Known hypersensitivity to the following drugs or constituents (and its excipients): methylprednisolone, prednisone, upadacitinib, or upadacitinib placebo. The following ingredients can be found in upadacitinib and upadacitinib placebo: colloidal silicon dioxide, hypromellose, iron oxide yellow and iron oxide red, magnesium stearate, mannitol, microcrystalline cellulose, polyvinyl alcohol, polyethylene glycol, talc, tartaric acid and titanium dioxide. This includes a known or suspected hypersensitivity to cow's milk for patients expected to be in the inpatient cohort (component of methylprednisolone).
* Participants that are currently pregnant or breastfeeding. Participants with a borderline serum pregnancy test at Screening must have absence of clinical suspicion of pregnancy or other pathological causes of borderline results and a serum pregnancy test ≥ 3 days later to document continued lack of a positive result. Participants with a urine pregnancy test at Baseline that is borderline or ambiguous must have a serum pregnancy test performed. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive.
* Participants that have received any live vaccine with replicating potential within 30 days prior to the first dose of study drug or are expected to need a live vaccination with any replicating potential during study participation or within 30 days of study completion.
* Patients that meet diagnostic criteria for toxic megacolon as determined by the study and treatment team. Patients are expected to have dilation of the transverse colon > 6 centimeters (cm) or cecum/right colon > 9cm and three of the following signs of systemic toxicity (Temperature > 38◦C, Heart rate (HR) > 120 beats per minute (BPM), white blood cells (WBC) > 10500/microliter (µL), Hemoglobin < 10.5mg/dL) and one of the following (dehydration, altered mental status, severe electrolyte disturbances, or hypotension)
* Patients with active Cytomegalovirus (CMV) colitis as defined as having > 5 CMV inclusion bodies per high powered field in any one ulcer at baseline. If CMV colitis is confirmed, the patient can remain in the trial if permissible by the infectious disease and primary treatment team and if concomitant anti-viral therapy is initiated.
* Patients that had received any investigational agent or procedure within 30 days or five half-lives prior to baseline, whichever is longer, or were enrolled in an interventional study.
* Patients with an active malignancy with the exception of non-metastatic basal cell or squamous cell carcinoma of the skin or localized carcinoma in situ of the cervix.
* Patients that had a history of colectomy (total or subtotal), ileoanal pouch, Kock pouch, or ileostomy or were planning bowel surgery (partial colectomy is permissible)
* Patients with certain laboratory abnormalities suggestive of moderate or severe renal, hematological, or gastrointestinal/liver impairment (per protocol).
* History of or clinical evidence of liver cirrhosis
* History of inherited or acquired conditions that predispose to hypercoagulability (per protocol). Please note, that patients with a remote history of provoked thromboembolic event or recent thromboembolic event on systemic anticoagulation are NOT exclusionary.
* Active Hepatitis B Infection: Hepatitis B surface antigen (HBsAg) positive with detectable deoxyribonucleic acid (DNA) not on therapy. Patients with serologic evidence of a resolved prior hepatitis B virus (HBV) infection (i.e., HBsAg-negative and anti-HB Core-positive) or patients with HBsAg positive on suppressive HBV therapy with low DNA (<105 copies/milliliter (mL) or <104 IU/mL negative) are not exclusionary.
* Active Hepatitis C Infection: Hepatitis C Virus (HCV) ribonucleic acid detectable in any patient with anti-HCV antibody.
* Acquired Immunodeficiency Syndrome: Confirmed positive anti-human immunodeficiency virus (HIV) antibody with cluster of differentiation 4 (CD4) counts <350 cells/microliter (uL) or Acquired Immune Deficiency Syndrome (AIDS)- defining opportunist infection.
* Solid organ or bone marrow transplant within 1 year or expected transplant within 6 months of randomization.
* Patients that had a history of spontaneous GI perforation (other than appendicitis or mechanical injury) or are at significantly increased risk of GI perforation per investigator's judgment.
* Actively receiving strong CYP3A4 inducers or inhibitors prior to the first dose of study drug or are expected to receive any of these medications during the study period. This includes grapefruit and grapefruit juice.
* The presence of any condition possibly affecting oral drug absorption (e.g., gastrectomy, clinically significant diabetic gastroenteropathy, or certain types of bariatric surgery) as determined by the investigator. Procedures such as gastric banding that simply divide the stomach into separate chambers are not exclusionary.
* Patients that had a history of a clinically significant medical condition per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-01-16 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with an initial clinical response without rescue therapy or colectomy by treatment Day 5 after initiating induction therapy in the upadacitinib and corticosteroid arm compared to the corticosteroid monotherapy arm | Treatment 5 days
  Initial Clinical Response Definition:
  * A reduction in liquid bowel movements per 24 hours by ≥ 60% from randomization AND a C-reactive protein (CRP) < 1.5 milligrams per deciliter (mg/dL) AND no more than trace blood in stool, or
  * 4 liquid bowel movements or less per 24 hours AND a C-reactive protein (CRP) < 1.5 mg/dL AND no more than trace blood in stool.
  Liquid bowel movements are defined as completely liquid (Bristol stool chart type 7) or mostly liquid (Bristol stool chart type 8).
  If the patient is discharged prior to outcome assessment on treatment Day 5, the most recent CRP prior to treatment Day 5 will be to evaluate primary outcome (carry forward manner). If a patient has not experienced CRP improvement to <1.5mg/dL prior to discharge, patient will be requested to obtain a treatment Day 5 CRP as an outpatient lab on treatment Day 5.

SECONDARY OUTCOMES:
The proportion of participants in the outpatient cohort with a hospital admission by end of the acute induction phase (Day 5) in the upadacitinib and corticosteroid arm compared to the corticosteroid monotherapy arm. | Day 5
The proportion of participants undergoing colectomy without rescue therapy by the end of the post-acute induction phase (week 8/day 56) in the upadacitinib and corticosteroid arm compared to the corticosteroid monotherapy arm | Week 8 (day 56)
The proportion of participants undergoing colectomy without rescue therapy by week 12/Day 84 in the upadacitinib and corticosteroid arm compared to the corticosteroid monotherapy arm | Week 12 (Day 84)
The proportion of participants undergoing colectomy without rescue therapy by Week 48/Day 336 in the upadacitinib and corticosteroid arm compared to the corticosteroid monotherapy arm | Week 48 (Day 336)
The proportion of participants in clinical response without colectomy or rescue therapy by end of post-acute induction phase (week 8/day 56) in the upadacitinib and corticosteroid arm compared corticosteroid monotherapy arm | Week 8 (day 56)
  Clinical response is defined by having a C-reactive protein (CRP) <0.8 mg/dL AND ≤ 4 liquid bowel movements per 24 hours and no more than trace blood in stool.
The proportion of participants in clinical response without colectomy or rescue therapy by week 12/Day 84 in the upadacitinib and corticosteroid arm compared corticosteroid monotherapy arm | Week 12 (Day 84)
  Clinical response is defined by having a C-reactive protein (CRP) <0.8 mg/dL AND ≤ 4 liquid bowel movements per 24 hours and no more than trace blood in stool.
The proportion of participants in clinical response without colectomy or rescue therapy by week 48/Day 336 in the upadacitinib and corticosteroid arm compared corticosteroid monotherapy arm | Week 48 (Day 336)
  Clinical response is defined by having a C-reactive protein (CRP) <0.8 mg/dL AND ≤ 4 liquid bowel movements per 24 hours and no more than trace blood in stool.
The proportion of participants in corticosteroid-free clinical remission without colectomy or rescue therapy by week 8/Day 56 in the upadacitinib and corticosteroid compared to corticosteroid monotherapy arm | Week 8 (Day 56)
  Clinical remission is defined as having ≤ 2 liquid bowel movements per 24 hours and having visible rectal bleeding score of 0. Corticosteroid-free clinical remission is defined as being in clinical remission without the use of corticosteroids ≥ 14 days prior to time-point
The proportion of participants in corticosteroid-free clinical remission without colectomy or rescue therapy by week 12/Day 84 in the upadacitinib and corticosteroid compared to corticosteroid monotherapy arm | Week 12 (Day 84)
  Clinical remission is defined as having ≤ 2 liquid bowel movements per 24 hours and having visible rectal bleeding score of 0. Corticosteroid-free clinical remission is defined as being in clinical remission without the use of corticosteroids ≥ 14 days prior to time-point
The proportion of participants in corticosteroid-free clinical remission without colectomy or rescue therapy by week 48/Day 336 in the upadacitinib and corticosteroid compared to corticosteroid monotherapy arm | Week 48 (Day 336)
  Clinical remission is defined as having ≤ 2 liquid bowel movements per 24 hours and having visible rectal bleeding score of 0. Corticosteroid-free clinical remission is defined as being in clinical remission without the use of corticosteroids ≥ 14 days prior to time-point
Incidence and severity of adverse events by end of the Acute Induction Phase (Inpatient Cohort: 0-10 days; Outpatient Cohort: 5 days) | End of the acute induction phase (0-10 days) in the safety population
  Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence and severity of adverse events by the end of the post-acute induction phase (week 8/Day 56) | Post-acute induction phase (week 8/Day 56) in the safety population
  Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence and severity of adverse events by week 12/Day 84 | Week 12 (Day 84) in the safety population
  Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence and severity of adverse events by week 52/Day 365 (Study period + 4-week safety follow-up period) in the safety population | Week 52 (Day 365) in the safety population
  Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence of serious infections by end of the acute induction phase (0-10 days) | Acute induction phase (0-10 days) in the safety population
  Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence of serious infections by post-acute induction phase week 8/Day 56 | Week 8 (Day 56) in the safety population
  Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence of serious infections by end of week 12/Day 84 | Week 12 (Day 84) in the safety population
  Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence of serious infections by Week 52/Day 365 (Study Period + 4-week Safety Follow-up) | Week 52 (Day 365) in the safety population
  Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence and severity of adverse events of special interest (AESI) by end of the acute induction phase (0-10 days) | Acute induction phase (0-10 days) in the safety population
  Adverse events of special interest include serious infections, opportunistic infections, herpes zoster, active TB, malignancy (all types), adjudicated gastrointestinal perforations, adjudicated cardiovascular events (e.g., major adverse cardiac event (MACE)), anemia, neutropenia, lymphopenia, renal dysfunction, hepatic disorder, adjudicated embolic and thrombotic events (non-cardiac, non-central nervous system), serious hypersensitivity reactions, bone fracture, and retinal detachment. Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence and severity of adverse events of special interest by week 8/Day 56 | Week 8 (Day 56) in the safety population
  Adverse events of special interest include serious infections, opportunistic infections, herpes zoster, active TB, malignancy (all types), adjudicated gastrointestinal perforations, adjudicated cardiovascular events (e.g., major adverse cardiac event (MACE)), anemia, neutropenia, lymphopenia, renal dysfunction, hepatic disorder, adjudicated embolic and thrombotic events (non-cardiac, non-central nervous system), serious hypersensitivity reactions, bone fracture, and retinal detachment. Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence and severity of adverse events of special interest by week 12/Day 84 | Week 12 (Day 84) in the safety population.
  Adverse events of special interest include serious infections, opportunistic infections, herpes zoster, active TB, malignancy (all types), adjudicated gastrointestinal perforations, adjudicated cardiovascular events (e.g., major adverse cardiac event (MACE)), anemia, neutropenia, lymphopenia, renal dysfunction, hepatic disorder, adjudicated embolic and thrombotic events (non-cardiac, non-central nervous system), serious hypersensitivity reactions, bone fracture, and retinal detachment. Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug
Incidence and severity of adverse events of special interest for by week 52/Day 365 (Study period + 4-week Safety Follow-up Period) in the safety population | Week 52 (Day 365) in the safety population.
  Adverse events of special interest include serious infections, opportunistic infections, herpes zoster, active TB, malignancy (all types), adjudicated gastrointestinal perforations, adjudicated cardiovascular events (e.g., major adverse cardiac event (MACE)), anemia, neutropenia, lymphopenia, renal dysfunction, hepatic disorder, adjudicated embolic and thrombotic events (non-cardiac, non-central nervous system), serious hypersensitivity reactions, bone fracture, and retinal detachment. Adverse events will be graded to the 5 criteria as described in the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) v5.
  Safety population includes all participants that received at least one dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Berinstein, MD, MSc, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No